CLINICAL TRIAL: NCT04202484
Title: A Prospective, Single-arm, Exploratory Clinical Research on the Efficacy and Safety of Tripletrumab Combined With Oxaliplatin and Teggio (SOX) in First-line Treatment of Unresectable Locally Advanced or Metastatic Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Tripletrumab Combined With Oxaliplatin and Teggio (SOX) in First-line Treatment of Gastric and Gastroesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLK-XXY-1
Record Dates: First submitted 2019-12-05; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Gastric Cancer
Keywords: Immunotherapy; Efficacy; Safety
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Tegafur; gimeracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab combine CT (Experimental)
  Interventions: Drug: Toripalimab combined with oxaliplatin and Tegafur,Gimeracil and Oteracil Porassium Capsules

INTERVENTIONS:
Drug: Toripalimab combined with oxaliplatin and Tegafur,Gimeracil and Oteracil Porassium Capsules — Toripalimab: 240mg IV Q3W;Tegafur,Gimeracil and Oteracil Porassium Capsules: 40mg/m2 Bid PO×14d Q3W;Oxaliplatin: 130mg/m2 IV Q3W

SUMMARY:
The aim population is histopathologically confirmed locally unresectable advanced recurrent or metastatic adenocarcinoma of the gastric and gastroesophageal junction. Purpose of research to evaluate the efficacy and safety of tripletrumab combined with oxaliplatin and teggio (SOX) in first-line treatment of unreactable locally advanced, recurrent or metastatic gastric and gastroesophageal junction adenocarcinoma.

Every 21 days is a cycle, and treatment is scheduled for 6 cycles. Chemotherapy drugs until disease progression, toxicity intolerance, the start of new anti - tumor treatment, withdrawal, loss of access or death, etc., already reached first, shall be the basis for termination.

Treatment was effective for more than 6 treatment cycles and toxicity was, the subjects were judged by the researchers when to terminate the treatment and adjust the follow-up treatment plan.

For disease progression, toxicity intolerance, and initiation of new antitumor therapies.

For subjects who donot reach terminal events such as treatment, withdrawal, loss of follow-up or death, at the end of chemotherapy , the follow-up maintenance regimen was adjusted according to the researchers' evaluation.

The screening period of the study was 14 days. The screening test was completed and the evaluation was completed.

Subjects with standard discharge entered the treatment period, and the frequency of administration was determined according to the protocol.

Conduct treatment and complete relevant tests and assessments before each administration.

Tumor imaging was assessed every 6 weeks (±7 days) and all subjects were treated.

At the end of the visit, safety and imaging evaluations should be completed. Complete follow-up was conducted for a total of 90 days. Continue to receive tumor evaluation and imaging at a frequency of 2-3 months. Evaluation until disease progression, new antitumor therapy, withdrawal, Lost or dead, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80;
2. Radiographic findings were consistent with non-resectable locally advanced, recurrent or metastatic gastric and gastroesophageal junction adenocarcinoma;
3. Non-resectable locally advanced, recurrent or metastatic adenocarcinoma of the gastric and gastroesophageal junction (including sig-ring cell carcinoma and adhesion) confirmed by histopathological examination Liquid adenocarcinoma, hepatoid adenocarcinoma);
4. ECOG 0-1;
5. Adequate organ and bone marrow function, as defined below:

1) blood routine examination: absolute neutrophil count (ANC) ≥1.5×109/L; platelet count (PLT) ≥85×109/L; hemoglobin (HGB) 90 g/L or higher; 2) liver function: total bilirubin (TBIL) ≤2× normal upper limit (ULN) was required in patients without liver metastasis; alanine aminotransferase (ALT) and amino transferase (AST) ≤2.5×ULN.Requirements for patients with liver metastasis: serum total bilirubin (TBIL) ≤2× normal upper limit (ULN); alanine ammonia ALT and AST were ≤5×ULN; 3) renal function: creatinine clearance rate (Ccr) ≥60mL/min; 4) full coagulation function, defined as the international standardized ratio (INR) or prothrombin time (PT) ≤1.5 ULN; 6. According to RECIST v1.1, there is at least one measurable lesion or evaluable lesion; 7. Previous (new) adjuvant chemotherapy/adjuvant radiotherapy ending time to disease recurrence time >6 months; 8. Expected survival time ≥12 weeks; 9. Female subjects of child-bearing age or male subjects whose sexual partners are female of child-bearing age shall take effective contraception throughout the treatment period and 6 months after the treatment period measures; 10. Subjects voluntarily participate in the study, sign the informed consent, and comply with the protocol visit and related procedures.

Exclusion Criteria:

1. Adenocarcinoma of the gastric and gastroesophageal junction diagnosed as HER2 positive; Previous exposure to any anti-pd-1 or anti-pd-l1, pd-l2, CD137, ctla-4 antibody therapy, or any other antibodies or drugs specifically targeting T cell co-stimulation or checkpoint pathways; Previous systematic treatment for advanced or metastatic adenocarcinoma of the gastric and gastroesophageal junction;
2. Participate in another interventional clinical study, unless participating in an observational (non-interventional) clinical study or in the follow-up phase of the interventional study;
3. Patients with autoimmune diseases or abnormal immune system;
4. The history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation is known; uncontrolled high blood pressure, diabetes and heart disease;
5. Cardia and pylorus are nearly obstructed, affecting the patient's eating and stomach emptying, or swallowing tablets is obstructed; The signs of lesion activity bleeding under endoscopy are known;
6. Known active tuberculosis; Interstitial lung disease requiring steroid ormone therapy;
7. A known history of human immunodeficiency virus (HIV) infection (i.e. HIV antibody positive); Acute or chronic active hepatitis b (HBsAg positive with HBV DNA viral load ≥200 IU/mL or ≥103 copy number /mL) or acute or chronic active hepatitis c (HCV antibody positive and HCV RNA positive) is known.
8. Severe infections in the active phase or poorly controlled clinically;
9. History of other primary malignant tumors, except: malignant tumors that had been in complete remission for at least 2 years before enrollment and did not require other treatment during the study period; Non-melanoma skin cancer or malignant freckle mole with adequate treatment and no evidence of disease recurrence; Carcinoma in situ with adequate treatment and no evidence of disease recurrence;
10. Female patients who are pregnant or breastfeeding;
11. Known allergy to any monoclonal antibody or component of the preparation of chemotherapy drugs (teggio, oxaliplatin) (grade 3 or higher);
12. Clinically significant ascites, including any ascites that can be found on physical examination, ascites that have been previously treated or are still in need of treatment, with only a small amount of ascites shown on imaging but no symptoms, can be included. Patients with bilateral medium pleural effusion, or large pleural effusion, or respiratory dysfunction requiring drainage;
13. Other acute or chronic diseases, mental illnesses, or laboratory abnormalities that may result in increased risk of study participation or study drug administration, or interfere with the interpretation of the study results, and in the judgment of the investigator, the patient is not eligible to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | All subjects receive tumor assessment every 6 weeks until desease progress, up to 24mons. Objective response rate is defined as the date from ICF signation to the date of first documented progression or date of death from any cause, whichever came first.
  The percentage of patients whose tumors shrink to a certain extent and remain there for a certain period of time, including CR+PR cases

IPD SHARING:
Plan to Share IPD: No